CLINICAL TRIAL: NCT07387614
Title: WEB-BASED SUPPORT PROGRAM FOR CAREGIVERS OF VETERANS WITH DEMENTIA DISCHARGED FROM SKILLED NURSING FACILITIES TO HOME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Molly Horstman, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-55864; 5P30AG086563-02 (NIH)
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Caregivers

STUDY DESIGN:
Intervention Model Description: This is an unblinded, parallel group, randomized trial of a 3-month caregiver support intervention (Hospital GamePlan4Care) for caregivers of hospitalized Veterans with dementia discharged to skilled nursing facilities compared to health education.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital GamePlan4Care (Experimental): Tailored caregiver skills training and support for caregiving for a person with dementia
  Interventions: Behavioral: Hospital GamePlan4Care
- Health Education (Active Comparator): Education on general caregiving topics.
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: Hospital GamePlan4Care — The Hospital GamePlan4Care intervention will include access to a written VA Care Transitions handbook, access to the GamePlan4Care website for skills training, 11 emails encouraging them to visit the website, and four phone calls with a dementia care specialist to tailor the training to the caregiver's needs over a 3-month period
  Arms: Hospital GamePlan4Care
Other: Health Education — Caregivers in the health education arm will receive a VA Care Transitions Handbook, 4 emails with a weblink to a general caregiving topic, and 4 phone calls to confirm that the emails were received over a 3-month period.
  Arms: Health Education

SUMMARY:
The goal of this clinical trial is to learn whether an evidence-based caregiver support program (Hospital GamePlan4Care) can benefit caregivers of hospitalized Veterans with Alzheimer's Disease and Related Dementia who are discharged to skilled nursing facilities prior to returning home. The main questions it aims to answer are:

* Is Hospital GamePlan4Care feasible and acceptable to caregivers?
* Does Hospital GamePlan4Care improve caregiver-reported outcomes?

Researchers will compare Hospital GamePlan4Care to health education to see if it improves caregiver reported outcomes.

Participants in the Hospital GamePlan4Care arm will receive tailored skills training and support. Participants will be asked to:

* Complete tailored skills training on the Hospital GamePlan4Care website
* Complete four phone calls with a dementia care specialist to receive tailored training and support
* Complete questionnaires at enrollment, one month, and three months after enrollment.
* Complete an interview at three months

Participants in the health education arm will receive education materials for caregivers. Participants will be asked to:

* Review the education materials
* Complete four phone calls with a dementia care specialist to review the materials
* Complete questionnaires at enrollment, one month, and three months after enrollment.

DETAILED DESCRIPTION:
Hospital GamePlan4Care is an evidence-informed intervention designed to support caregivers of hospitalized adults with dementia. Hospital GamePlan4Care was developed and tested with feedback from caregivers and health professionals and found to be feasible and acceptable to caregivers in a single arm pilot study. Hospitalization of an adult with dementia can be associated with negative outcomes for the adult with dementia (e.g., cognitive decline, functional decline) and caregivers (e.g., depression, increased stress), which may place the adult with dementia at increased risk for elder mistreatment following hospital discharge. Supporting caregivers during care transitions may improve outcomes for caregivers and mediate the risk for elder mistreatment. This clinical trial addresses an important gap in our understanding of the potential benefits of caregiver-support programs during care transitions for caregivers and adults with dementia.

This study will be a non-blinded randomized study comparing Hospital GamePlan4Care (intervention arm) to a Health Education (control arm) for caregivers of hospitalized Veterans with dementia who are discharged to a skilled nursing facility prior to returning home. Caregivers of adults with dementia will be recruited while the Veteran is admitted to a skilled nursing facility after hospital discharge. Following baseline data collection, enrolled caregivers will be randomized to Hospital GamePlan4Care or Caregiver Education arm in a 1:1 ratio using the randomization feature in VA REDCap. Each arm will continue for three months after the caregiver is enrolled. The primary outcomes are caregiver-reported and will be measured 30 days and 90 days after caregiver enrollment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* provide care for a Veteran with a diagnosis of Alzheimer's Disease or related dementias or a Veteran with a prescription for a medication for dementia listed in CPRS who is admitted to the hospital at the Michael E. DeBakey VA Medical Center
* Veteran must be experiencing signs of dementia as verified by a score of 2 or greater on the AD-8
* care for a Veteran with dementia who is discharged to a VA or non-VA skilled nursing facility prior to returning home
* provide at least eight hours of care or supervision per week to the Veteran with dementia
* provide care primarily due to a personal relationship, rather than a financial relationship
* have access to a telephone
* have access to a tablet or computer with internet access
* report using the computer or tablet to access the internet at least three times per week
* speak English

Exclusion Criteria:

* unable to complete informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2027-02-17 (Estimated); Study Completion 2027-02-17 (Estimated)

PRIMARY OUTCOMES:
Caregiver Unmet Needs: Benjamin Rose Unmet Needs Scale | Baseline, 30 days and 90 days
  The Benjamin Rose Institute Unmet Need Scale includes 39 yes/no questions about different need that caregivers have (no=0, yes=1). The total score is a sum of all the yes responses. Higher scores indicate higher unmet needs.

SECONDARY OUTCOMES:
Change in Self-Efficacy for Caregiving (CSES-8) | Baseline, 30 days, and 90 days
  The CSES-8 asks questions about confidence in being able to manage different caregiving situations. Each question is rated on a 1 (not at all confident) to 10 (totally confident scale). The score of the scale is the mean of the eight items. Higher scores indicate greater self-efficacy.
Change in Center for Epidemiological Studies Depression Scale (CES-D) (10-item) | Baseline, 30 days, and 90 days
  The CES-D provides a list of feelings and behaviors. For each item, respondents report how often they have felt that way in the past week with each item receiving a score from 0-3. A total score will be obtained by summing scores for all items with higher scores indicating higher levels of depressed symptoms (range: 0-30).
Change in Zarit Caregiving Burden Interview (12-item) | Baseline, 30 days and 90 days
  Each item represents a statement related to an aspect of perceived burden. All questions are answered as never (0 points), rarely (1 point), sometimes (2 points), quite frequently (3 points), or nearly always (4 points). A total score will be obtained by summing all items with higher scores indicating higher rates of burden (range: 0-48).
Change in Self-Rated Health (1-item) | Baseline, 30 days, and 90 days
  The investigators will use the single self-rated health item: "In general, would you say your health is:" with response options of Excellent, Very Good, Good, Fair, and Poor
Change in Caregiver Distress on the Neuropsychiatric Inventory Questionnaire | Baseline, 30 days, and 90 days
  The Neuropsychiatric Inventory Questionnaire includes a list of 12 symptoms (e.g. delusions, hallucinations, agitation/aggression). For each symptom, the caregiver responds if the symptom was present in the past month (yes/no) and the level of distress the caregiver feels due to that symptom (0-5). Higher scores indicate greater distress due to that symptom.
Neglect and Aggression Questionnaire | Baseline, 30 days, and 90 days
  Questions adapted from the Conflict Tactics Scale Revised and CTS2 modified for older adults; Conflict Tactics Scale for Child Mistreatment; and prior research (Pickering 2024, PMID 39136354). Asks how often the caregiver or care recipient has done I something in the past month. Questions include neglect of the care recipient, caregiver self-neglect, physical and psychological aggression of the caregiver to the care recipient, and physical and psychological aggression of the care recipient to the caregiver.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide a de-identified dataset compliant with VA data security policy to the public upon request to the principal investigator.
Time Frame: After the data is analyzed and published